CLINICAL TRIAL: NCT02711163
Title: Evaluation of the Hypoallergenicity of a New Thickened Extensively Hydrolyzed Formula in Infants With Confirmed Cow's Milk Protein Allergy
Brief Title: Evaluation of the Hypoallergenicity of an Extensively Hydrolyzed Formula
Acronym: ALYCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UP-2014-02-ALYCE
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extensively hydrolyzed formula (Experimental): Feeding extensively hydrolyzed formula
  Interventions: Dietary Supplement: Extensively Hydrolyzed formula
- Amino acid formula (Placebo Comparator): Feeding amino acid formula
  Interventions: Dietary Supplement: Amino acid formula

INTERVENTIONS:
Dietary Supplement: Extensively Hydrolyzed formula
  Arms: Extensively hydrolyzed formula
Dietary Supplement: Amino acid formula
  Arms: Amino acid formula

SUMMARY:
The aim of this study is to assess the hypoallergenicity of a new thickened extensively hydrolyzed formula, in infants with confirmed cow's milk protein allergy assessed through a double blind placebo controlled food challenge, followed by a 3-month open feeding period.

ELIGIBILITY:
Main Inclusion Criteria:

Infants:

* with cow's milk allergy confirmed by a double-blind food challenge performed in the last 2 months,
* successfully fed an eviction diet for at least 2 weeks

Main Non-inclusion Criteria:

Infants:

* fed with an extensively hydrolyzed formula with no improvement of the symptoms,
* who refused to drink an extensively hydrolyzed formula anytime prior to inclusion,
* fed a vegetable based formula
* fed an amino acid based formula or who should be fed with an amino acid based formula according to recommendations
* who had an anaphylactic reaction in the past

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08-31 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Percentage of infants tolerating the formula during a double blind placebo controlled food challenge | 7 days

SECONDARY OUTCOMES:
Regurgitation assessed through Vandenplas score | 7, 45 and 90 days
Vomiting (weekly frequency) | 7, 45 and 90 days
Abdominal pain (severity on a 4 level scale) | 7, 45 and 90 days
Bloating and gas (severity on a 4 level scale) | 7, 45 and 90 days
Stool consistency assessed through Bristol Stools Form Scale | 7, 45 and 90 days
Sleeping time over 24h | 7, 45 and 90 days
Stool frequency over 72h | 7, 45 and 90 days
Blood in stools (presence/absence) | 7, 45 and 90 days
Duration of crying over 24h | 7, 45 and 90 days
Respiratory symptoms (severity on a 4 level scale) | 7, 45 and 90 days
Urticaria (presence/absence) | 7, 45 and 90 days
Eczema assessed through SCORAD | 7, 45 and 90 days
Weight expressed in z scores according to the WHO Child Growth Standards | 45 and 90 days
Height expressed in z scores according to the WHO Child Growth Standards | 45 and 90 days
BMI expressed in z scores according to the WHO Child Growth Standards | 45 and 90 days
Head circumference expressed in z scores according to the WHO Child Growth Standards | 45 and 90 days
Number of patients with treatment emergent Adverse Events | 7, 45 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Cucchiara, Principal Investigator — University Hospital Umberto I
Locations (1):
- Umberto I university hospital, Roma, Italy